CLINICAL TRIAL: NCT05752643
Title: Feasibility and Impact of Online HIV/STI Screening Addressed to Men Who Have Sex With Men and Transgender Women Pre-exposure Prophylaxis (PrEP) Users in Spain
Brief Title: Feasibility and Impact of Online HIV/STI Screening Addressed to PrEP Users in Spain
Acronym: TESTATE_PrEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Collaborators: Department of Health, Generalitat de Catalunya (Other Government); Hospital Vall d'Hebron (Other)
Responsible Party: Principal Investigator, Cristina Agusti, Principal Investigator, Fundació Institut Germans Trias i Pujol
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CEEISCATTESTATEPrEP
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: HIV; STI
Keywords: HIV; STI; Pre-exposure prophylaxis (PrEP); e-STI; Self-sampling; Screening; ICT
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: Non-blinded randomized controlled non-inferiority trial
Masking Description: Due to the nature of the intervention, participants will know to which arm they have been allocated. So, it would not be possible to blind either the participants or healthcare professionals
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will have 4 face-to-face quarterly follow up visits per year
- Experimental (Experimental): Participants will alternate face-to-face visits with online screening every three months. They will have two face-to-face and two online screenings per year
  Interventions: Other: Online follow up

INTERVENTIONS:
Other: Online follow up — The online follow up will include screening for HIV and STIs (Chlamydia trachomatis (CT), Neisseria gonorrhoeae (NG) and Treponema pallidum (TP)) based in a self-sampling strategy
  Arms: Experimental

SUMMARY:
Non-blinded randomized controlled non-inferiority trial to evaluate the feasibility, acceptability and impact of an innovative internet-accessed HIV and STIs screening intervention (TÉSTATE PrEP) addressed to gays, bisexuals and other men who have sex with men (GBMSM) and transgender women users of PrEP in Spain as part of PrEP follow up.

DETAILED DESCRIPTION:
The objectives of the study are 1) To design and implement an e-HIV/STI testing pilot intervention (TÉSTATE PrEP) to offer self-sampling kits to detect HIV, Chlamydia trachomatis (CT), Neisseria gonorrhoeae (NG) and Treponema pallidum (TP) among gays, bisexuals and other men who have sex with men (GBMSM) and transgender women users of pre-exposure prophylaxis (PrEP) as part of PrEP follow up. 2) To evaluate if the pilot does not cause a reduction of the retention to PrEP follow up among the target population. 3) To analyze the capacity of the intervention to reduce the healthcare burden of the PrEP service. 4) To evaluate the acceptability of the intervention among PrEP users and healthcare workers of the PrEP services; and 5) To validate dried blood samples (DBS) for confirmation of TP infection and performing RPR to determine stage and activity of infection comparing with blood drawn by venous puncture. Investigators will perform a non-blinded randomized controlled non-inferiority trial among PrEP users on follow up in one of the main PrEP services of Spain. Participants on the control arm will follow the usual follow up protocol with quarterly face-to-face visits where they will be tested for HIV and STIs. Participants in the experimental arm will alternate face-to-face meetings with online screening of HIV and STIs. This project is based on the TÉSTATE project (PI17 00355). The website https://testate.org/ will include a module for online follow-up visits of participants on PrEP. Participants of the experimental arm will register in the website and will receive self-sampling kits to their home to get tested for HIV, CT, NG and TP. Participants will send the samples to the reference laboratory and check their results online. The investigators will compare the retention to follow up among PrEP users in the control and experimental arm and the healthcare burden in each group. The acceptability of the intervention among the PrEP users and healthcare workers will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* GBMSM or transgender women
* PrEP users with more than 1 year of follow up in the collaborating center (The Centre for International Health and Infectious Diseases Drassanes Vall d'Hebron (Barcelona))
* Not having altered renal function
* Resident in Spain

Exclusion Criteria:

* Not able to read in Spanish
* Not able to give their consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender Men who are gay, bisexual and other men who have sex with men (GBMSM) ; and Transgender women
Enrollment: 218 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Retention to PrEP follow up | Two years follow-up (from baseline to year 2)
  Proportion of PrEP users that who have not missed any follow-up visit: Number of participants who have not missed a follow up visit /total number of participants in follow up for PrEPx100 (%)
Healthcare burden | Two years follow-up (from baseline to year 2)
  Median number of visits per participant and year at the PrEP Service

SECONDARY OUTCOMES:
Proportion of participants diagnosed with HIV | Two years follow-up (from baseline to year 2)
  Proportion of participants diagnosed with HIV in each arm
Proportion of participants diagnosed with CT, NG and TP | Two years follow-up (from baseline to year 2)
  Proportion of participants diagnosed with CT, NG and TP infections in each arm
Proportion of participants who are prescribed treatment for HIV/STI | Two years follow-up (from baseline to year 2)
  Proportion of participants who are prescribed treatment for HIV/STI in each arm
Aherence to PrEP | Two years follow-up (from baseline to year 2)
  Aherence to PrEP in each arm
Samples sent to lab and results consulted | Two years follow-up (from baseline to year 2)
  Number of participants of the experimental arm who send the samples to the laboratory, and consult the results
Participants acceptability | Two years follow-up (from baseline to year 2)
  The proportion of participants in the intervention group who agree that the online follow up combined with the face-to-face follow up at the PrEP service is acceptable
Health professionals acceptability | Two years follow-up (from baseline to year 2)
  The proportion of health care professionals of the PrEP service who agree that the online follow up combined with the face-to-face follow up at the PrEP service is acceptable

IPD SHARING:
Plan to Share IPD: No
Only researchers in the study will be able to access this IPD. No data transfer will be made to third parties

REFERENCES:
- [Derived] Agusti C, Martinez Riveros H, Garcia-Perez J, Descalzo V, Fernandez G, Ramirez-Marinero A, Gonzalez MV, Diaz Y, Montoro-Fernandez M, Romano-deGea P, Araujo SG, Muntada E, Casabona J. Feasibility and impact of online HIV/STI screening addressed to men who have sex with men and transgender women users of pre-exposure prophylaxis (PrEP) in Spain (TESTATE PrEP): a study protocol for a non-blinded randomised controlled trial. BMJ Open. 2023 Oct 16;13(10):e073459. doi: 10.1136/bmjopen-2023-073459. PMID 37844988